CLINICAL TRIAL: NCT04452032
Title: Prospective Pilot Study Evaluating Dental Side Effects of Radiotherapy on Subjects Treated for Head and Neck Cancer
Acronym: StomRay
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IJB-RT-HNC-002
Record Dates: First submitted 2020-06-08; First posted 2020-06-30 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): The first phase of the study will consist of an evaluation of the initial dental state of each subject based on stomatological examination, orthopantomogram, bitewing radiographs, evaluation of potential risks of caries and fractures. Dental decalcification, dental care and/or avulsion if necessary, and afterwards, a dental splint will be performed before the start of RT treatment.Based on our predictive model, every tooth which potentially will receive more than 40 Gy and for which long term survival is compromised will be avulsed at least 2 weeks before the start of RT.
  After RT, the subject will have clinical follow-up with dental evaluation every 6 months for 36 months in order to identify possible dental events. At each consultation, a stomatological examination will be performed as well as bitewing radiographs. Orthopantomogram will be done once a year. Periapical X-rays will be performed if there is a dental complain or to refine a lesion visible on orthopantomogram.
  Interventions: Procedure: Dental avulsion; Radiation: Radiotherapy

INTERVENTIONS:
Procedure: Dental avulsion — Before radiotherapy, each subject undergoes a dental evaluation and if it is necessary, dental avulsions if their long-term survival is compromised (see in section 6.1.2) and if they are located in an area at risk to receive more than 40 Gy, so to develop osteoradionecrosis of the jaw. The avulsions should be performed as far as possible from the start of radiotherapy (RT) namely at least 2 weeks before irradiation to allow mucosal healing.
Radiation: Radiotherapy — Radiotherapy:
  All Subjects will be treated by simultaneous integrated boost (SIB) intensity modulated radiotherapy (IMRT) / volumetric modulated arc therapy (VMAT).

SUMMARY:
Multi-centric, one arm phase II study. The first phase of the study will consist of an evaluation of the initial dental state of each subject based on a stomatological examination, an orthopantomogram, two bitewing radiographs (right and left sides) and an evaluation of all potential risks of caries and fractures. For all of subjects, a dental decalcification, dental care and/or avulsion if necessary, and afterwards, a dental splint will be performed before the start of RT treatment. Our previously developed predictive model for dental dose in function of the localisation of tumour and suspect lymph nodes based on the stomatological examination and on the pre-treatment imaging. An estimation of the intensity-modulated radiotherapy (IMRT) teeth dose will be made and translated into a colour based form of the pre-RT dental status. A contouring of the teeth will be performed and the planned dose for each tooth of each subject will be recorded by a dose volume histogram (DVH) curve based on the pre-treatment imaging. In the same way the mean dose and the V25 (the volume receiving 25 Gy) of the homo- and the heterolateral parotid gland will be calculated. Based on our predictive model, every tooth which potentially will receive more than 40 Gy and for which long term survival is compromised will be avulsed at least 2 weeks before the start of RT.

After RT, the subject will have clinical follow-up with dental evaluation every 6 months for 36 months in order to identify possible dental events. At each consultation, a stomatological examination will be performed as well as two bitewing radiographs. An orthopantomogram will be done once a year. Furthermore, periapical X-rays will be performed if there is a dental complain or to refine a lesion visible on orthopantomogram.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. ECOG performance status ≤2
3. Female and Male
4. Newly diagnosed, histologically or cytologically confirmed head and neck squamous cell carcinoma (oropharynx, oral cavity, larynx, hypopharynx or cavum)
5. Results of previous pre-treatment imaging (PET-CT and cervicofacial MRI and/or CT/scan)
6. Eligible for treatment based on (chemo-)radiotherapy (with or without a surgical treatment)
7. Agree to wear, three times per week, fluoride dental splint after RT
8. HPV/p 16 testing results available at the time of screening (only for subjects with oropharynx cancer)
9. Serum pregnancy test (for subjects of childbearing potential) negative within 7 days prior to the 1st radiotherapy treatment
10. Women of childbearing potential must agree to use of one effective method of contraception prior study entry and during the course of the study.
11. Completion of all necessary screening procedures within 30 days prior to 1st radiotherapy treatment.
12. Signed Informed Consent form (ICF) obtained prior to any study related procedure.
13. Ability to understand and complete the questionnaires (language proficiency, cognitive functioning) as judged by the principal investigator upon screening

Note: Subject from the SwallPEG trial can participate in the StomRay study if they meet all of the previous eligibility criteria.

Exclusion Criteria:

1. Subject having less than ten teeth on dental arch
2. Life expectancy less than 12 months
3. History of previous head and neck irradiation
4. Prior or current treatment with bisphosphonates or denosumab
5. Presence of too many metal artefacts on the RT simulation scan preventing precise teeth contouring
6. Subject with a significant medical, neuro-psychiatric, or surgical condition, currently uncontrolled by treatment, which, in the principal investigator's opinion, may interfere with completion of the study.
7. Pregnancy and/or lactating women
8. Subjects with imperfect amelogenesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2026-05-16 (Estimated); Study Completion 2027-05-16 (Estimated)

PRIMARY OUTCOMES:
Risk of dental complication | At 36 months after end of radiotherapy
  Frequency of dental fractures according to the teeth radiotherapy delivered dose
Risk of dental complication | At 36 months after end of radiotherapy
  Frequency of dental caries according to the parotid radiotherapy delivered dose

SECONDARY OUTCOMES:
Validation of a "predictive dose model" of radiotherapy | At 36 months after end of radiotherapy
  Predictive dose of radiotherapy according to the location of the tumour
Validation of a "predictive dose model" of radiotherapy | At 36 months after end of radiotherapy
  Predictive dose of radiotherapy according to the TNM stage
Validation of a "predictive dose model" of radiotherapy | At 36 months after end of radiotherapy
  Predictive dose of radiotherapy with the real dose of radiotherapy received
Comparison of the predictive dose of radiotherapy with the dental complication probability | At 36 months after end of radiotherapy
  Number of dental caries per patient
Comparison of the predictive dose of radiotherapy with the dental complication probability | At 36 months after end of radiotherapy
  Number of dental fractures per patient
Comparison of the predictive dose of radiotherapy with the dental complication probability | At 36 months after end of radiotherapy
  Number of dental avulsions per patient
Assessment of Quality of life | At 36 months after end of radiotherapy
  Avulsion-free
Assessment of Quality of life | At 36 months after end of radiotherapy
  Number of patients who developp an osteoradionecrosis of the jaw
Assessment of Quality of life | At 36 months after end of radiotherapy
  Outcome measure: completion of xerostomia questionnaire
Assessment of Quality of life | At 36 months after end of radiotherapy
  Outcome measure: completion of EORTC: QLQ-C30 questionnaire
Assessment of Quality of life | At 36 months after end of radiotherapy
  Outcome measure: completion of EORTC: QLQ-H&N43 questionnaire

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - CHU saint Pierre, Brussels
  - Hôpital Erasme, Brussels
  - Institut Jules Bordet, Brussels